CLINICAL TRIAL: NCT06423612
Title: Randomized Trial to Optimize Virologic Suppression Rates Using a Point-of-Care Urine Monitoring Assay (ROVING PUMA)
Acronym: ROVING-PUMA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Desmond Tutu HIV Foundation (Other); University of Cape Town (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A143057; R01AI143340-06 (NIH)
Record Dates: First submitted 2024-05-16; First posted 2024-05-21 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: ART Adherence
Keywords: ART; Adherence; South Africa; Viral Suppression; ART resistance; POC urine assay; TDF assay

STUDY DESIGN:
Intervention Model Description: Randomized hybrid type 1 effectiveness trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- POC Urine Test Informed ART Adherence Counselling (Experimental): Conduct enhanced ART adherence counselling informed by the results of the point-of-care urine assay for TFV to increase viral suppression.
  Interventions: Behavioral: POC urine assay informed enhanced ART adherence counselling for viral suppression
- Standard-of-care Enhanced Adherence Counselling (No Intervention): Follow South Africa's standard-of-care enhanced ART adherence counselling for viral suppression.

INTERVENTIONS:
Behavioral: POC urine assay informed enhanced ART adherence counselling for viral suppression — Collect urine on intervention participants and screen for presence of TFV. Feedback will be provided to the participant based on the results on their ART adherence with provision of enhanced ART adherence counseling for viral suppression.
  Arms: POC Urine Test Informed ART Adherence Counselling

SUMMARY:
Antiretroviral therapy (ART) has significantly decreased the morbidity and mortality of HIV infection. However, adherence challenges in taking daily oral ART persist. A retrospective cohort study across 31 countries from 2010-19 reported that only 65% of people with HIV (PWH) on ART exhibited virologic suppression (VS) three years after starting ART;1 the rate of VS in South Africa among PWH on ART is 60-65%. Adherence barriers span individual and structural factors, such as stigma, recall difficulties, housing and/or food insecurity, mental illness, substance use, transportation, stock-outs, and other factors that vary by country and population.

Adherence interventions can benefit from direct objective adherence monitoring. Pharmacologic metrics of adherence assess drug levels in plasma, dried blood spots, hair (a metric our group pioneered) or urine and predict outcomes more accurately than self-reported adherence. However, most of these metrics preclude real-time assessment, requiring expensive laboratory equipment and trained laboratory personnel. Thus, few adherence interventions have successfully incorporated objective metrics, likely due to laboratory and shipping delays. A low-cost (<$2/test) point-of-care adherence metric - developed by our group - should allow for real-time biofeedback and improve the impact of metric-driven adherence interventions.

DETAILED DESCRIPTION:
This is a randomized hybrid type 1 effectiveness study design to assess the factors related to implementation of a point-of-care urine TFV assay test into routine HIV clinical care. We plan to recruit a total of 500 adults living with HIV who received primary HIV care from one of the selected study clinics in BCM, Eastern Cape. Individuals who have been prescribed ART for at least 6 months who have not achieved VS will be randomized in a 1:1 fashion at the baseline visit to the intervention arm vs. the SoC arm.

Total duration of the study is 18 months from the time of enrollment.

ELIGIBILITY:
Inclusion Criteria:

Aim 1: Individuals ≥18 years of age at the initial screening visit living with HIV, prescribed ART for at least three months, and are not virally suppressed.

Aim 2: Same as Aim 1 for the acceptability survey and in-depth interviews. HIV care providers in the selected clinic sites for the feasibility survey and in-depth interviews.

Aim 3: Same as Aim 1 for the cost-effectiveness study.

Exclusion Criteria:

* Currently enrolled in another ART adherence intervention
* Patients on ART regimen that does not include Tenofovir
* HIV care providers from non-study sites Failure to provide written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-05-08 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Viral Suppression at 6 months | 18 months
  The primary outcome of effectiveness will be viral suppression at 6 months.

SECONDARY OUTCOMES:
Viral suppression at 9, 12, and 18months | 18 months
  Durability of the 6-month intervention on viral suppression at 9, 12, and 18months
Resistance testing and genotype results @ 6 and 18 months | 18 months
  The effect of the intervention on need for resistance testing and genotype results @ 6 and 18 months
Feasibility and Acceptability of the intervention | 18 months
  Assess the feasibility and acceptability of the intervention using a survey and in-depth interviews
Cost-effectiveness of the intervention | 18 months
  Assess the cost per patient, cost per additional patient with VS, and cost per disability-adjusted life-year averted from a society perspective with using the urine-based TFV adherence assay to inform adherence counseling vs. standard of care counseling.

CONTACTS AND LOCATIONS:
Overall Officials: Monica Gandhi, Principal Investigator — University of California, San Francisco
Locations (1):
- Desmond Tutu HIV Foundation, East London, South Africa

IPD SHARING:
Plan to Share IPD: Yes
We will share de-identified data in publicly accessible databases once study is complete and study findings disseminated.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 48 months from start of study
Access Criteria: Investigators conducting ART adherence research.

REFERENCES:
- [Background] Niu X, Kubiak RW, Siriprakaisil O, Klinbuyaem V, Sukrakanchana PO, Cressey R, Okochi H, Gandhi M, Cressey TR, Drain PK. Tenofovir-Diphosphate in Dried Blood Spots vs Tenofovir in Urine/Plasma for Oral Preexposure Prophylaxis Adherence Monitoring. Open Forum Infect Dis. 2022 Aug 10;9(8):ofac405. doi: 10.1093/ofid/ofac405. eCollection 2022 Aug. PMID 36004315
- [Background] Spinelli MA, Haberer JE, Chai PR, Castillo-Mancilla J, Anderson PL, Gandhi M. Approaches to Objectively Measure Antiretroviral Medication Adherence and Drive Adherence Interventions. Curr HIV/AIDS Rep. 2020 Aug;17(4):301-314. doi: 10.1007/s11904-020-00502-5. PMID 32424549
- [Background] Gandhi M, Wang G, King R, Rodrigues WC, Vincent M, Glidden DV, Cressey TR, Bacchetti P, Spinelli MA, Okochi H, Siriprakaisil O, Klinbuayaem V, Mugo NR, Ngure K, Drain PK, Baeten JM. Development and validation of the first point-of-care assay to objectively monitor adherence to HIV treatment and prevention in real-time in routine settings. AIDS. 2020 Feb 1;34(2):255-260. doi: 10.1097/QAD.0000000000002395. PMID 31634188
- [Background] Cressey TR, Siriprakaisil O, Kubiak RW, Klinbuayaem V, Sukrakanchana PO, Quame-Amaglo J, Okochi H, Tawon Y, Cressey R, Baeten JM, Gandhi M, Drain PK. Plasma pharmacokinetics and urinary excretion of tenofovir following cessation in adults with controlled levels of adherence to tenofovir disoproxil fumarate. Int J Infect Dis. 2020 Aug;97:365-370. doi: 10.1016/j.ijid.2020.06.037. Epub 2020 Jun 14. PMID 32553717
- [Background] Drain PK, Bardon AR, Simoni JM, Cressey TR, Anderson P, Sevenler D, Olanrewaju AO, Gandhi M, Celum C. Point-of-care and Near Real-time Testing for Antiretroviral Adherence Monitoring to HIV Treatment and Prevention. Curr HIV/AIDS Rep. 2020 Oct;17(5):487-498. doi: 10.1007/s11904-020-00512-3. PMID 32627120
- [Background] Drain P, Ngure K, Mugo N, Spinelli M, Chatterjee P, Bacchetti P, Glidden D, Baeten J, Gandhi M. Testing a Real-Time Tenofovir Urine Adherence Assay for Monitoring and Providing Feedback to Preexposure Prophylaxis in Kenya (PUMA): Protocol for a Pilot Randomized Controlled Trial. JMIR Res Protoc. 2020 Apr 2;9(4):e15029. doi: 10.2196/15029. PMID 32238341